CLINICAL TRIAL: NCT07136610
Title: Standardized Application of Feeding Evaluations Using SMART Tool
Acronym: SAFEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00132685
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Infant and Young Child Feeding
Keywords: premature infants; medically complex infants; infant feeding; feeding skills assessment; length of stay; infant developmental assessment; dysphagia of newborn; cluster randomized trial; length of NICU stay; breastfeeding
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMART Tool (Experimental): Feeding skill assessment, the SMART Tool to monitor infant feeding skill development in the neonatal intensive care unit.
  Interventions: Behavioral: SMART Tool

INTERVENTIONS:
Behavioral: SMART Tool — The intervention in this implementation study involves (1) integrating the SMART Tool into electronic health records (EPIC), (2) educating all NICU staff (about 850 nurses, lactation consultants, speech-language pathologists, and physicians), and (3) Quality improvement to reinforce learning.
  Other Names: feeding skill assessment

SUMMARY:
Premature and medically complex infants have delayed development of oral feeding skills, leading to prolonged hospitalization, costs, and family stress. There is no "gold standard" infant feeding skill assessment tool for bedside clinicians. The research team developed a novel feeding skill assessment, the SMART Tool, to monitor infant feeding skill development in the neonatal intensive care unit. This study aims to determine whether this tool improves clinical outcomes, including reduced hospital days and enhanced safety and quality of infant feedings.

DETAILED DESCRIPTION:
The current recommendation for preventing infant feeding problems is to provide cue-based feeding, which entails optimizing feeding based on infant cues, including behavioral and physiological signs of stress. These recommendations rely on appropriately recognizing infant feeding cues to inform care instead of applying time-based, volume-driven care irrespective of cues. Care providers vary widely in their subjective assessment of feeding skills, often because they lack standard education on feeding skill assessment and a "gold standard" tool to objectively measure infant oral feeding skill levels. This robust, step-wedge, cluster randomized trial was designed to evaluate the effect of implementing the SMART Tool in 14 different Neonatal Intensive Care Units (NICU) in the Advocate Health Midwest Region. The SMART Tool is a novel feeding assessment tool developed at Advocate Illinois Masonic Medical Center to objectively measure feeding readiness and skill. The psychometric properties were tested through a research study, and strong validity and reliability were established. The Advocate Health Midwest Region NICU standardization committee approved this tool as the sole feeding skill assessment tool to be used at each oral feed (eight times a day) for all NICU infants. Data on infants in the NICU will abstracted from the medical record at the time of discharge or death. The study will use PRISM and the REAIM Framework. The implementation framework consists of three parts that interact to influence outcomes (contextual factors, roll-out strategies, outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Infants born between August 1, 2025, and July 31, 2026, AND admitted to NICU

Exclusion Criteria:

* No oral feeding started by July 15, 2026

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3500 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Month 6
  Days from birth to discharge
Number of days to full oral feeds | Month 6
  Days from birth to full oral feeds
Percent of Nasogastric tube days | Month 6
  Proportion of days with NG

SECONDARY OUTCOMES:
Home Tube Feeding | Month 6
  Proportion of infants discharged home with nasogastric tube or gastrosotomy tubes

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Mishra, MBBS, MD, Study Chair — Advocate Illinois Masonic Medical Center; Elizabeth Jensen, MPH, PhD, Principal Investigator — Wake Forest University Health Sciences; Joseph Chase, MPH, Principal Investigator — Advocate Aurora Research Institute; Anne Albi, BS, MS, Principal Investigator — Advocate Illinois Masonic Medical Center; Cynthia Lira-Crame, BSN, MSN, Principal Investigator — Advocate Illinois Masonic Medical Center
Locations (14):
- United States (14):
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Advocate Trinity Hospital, Chicago, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Advocate Condell Medical Center, Libertyville, Illinois
  - Advocate Christ Medical Center (Advocate Children's Hospital - Oak Lawn), Oak Lawn, Illinois
  - Advocate Lutheran General Hospital (Advocate Children's Hospital - Park Ridge), Park Ridge, Illinois
  - Aurora Medical Center Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Medical Center Kenosha, Kenosha, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Aurora Medical Center Oshkosh, Oshkosh, Wisconsin
  - Aurora Medical Center - Sheboygan County, Sheboygan, Wisconsin
  - Aurora Medical Center - Summit, Summit, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- [Background] Hemming K, Taljaard M. Key considerations for designing, conducting and analysing a cluster randomized trial. Int J Epidemiol. 2023 Oct 5;52(5):1648-1658. doi: 10.1093/ije/dyad064. PMID 37203433
- [Background] Glasgow RE, Trinkley KE, Ford B, Rabin BA. The Application and Evolution of the Practical, Robust Implementation and Sustainability Model (PRISM): History and Innovations. Glob Implement Res Appl. 2024;4(4):404-420. doi: 10.1007/s43477-024-00134-6. Epub 2024 Aug 31. PMID 39568619
- [Background] Browne JV, Jaeger CB, Kenner C; Gravens Consensus Committee on Infant and Family Centered Developmental Care. Executive summary: standards, competencies, and recommended best practices for infant- and family-centered developmental care in the intensive care unit. J Perinatol. 2020 Sep;40(Suppl 1):5-10. doi: 10.1038/s41372-020-0767-1. PMID 32859958
- [Background] Russ SA, Hotez E, Berghaus M, Verbiest S, Hoover C, Schor EL, Halfon N. What Makes an Intervention a Life Course Intervention? Pediatrics. 2022 May 1;149(Suppl 5):e2021053509D. doi: 10.1542/peds.2021-053509D. PMID 35503318
- [Background] Sanders MR, Hall SL. Trauma-informed care in the newborn intensive care unit: promoting safety, security and connectedness. J Perinatol. 2018 Jan;38(1):3-10. doi: 10.1038/jp.2017.124. Epub 2017 Aug 17. PMID 28817114
- [Background] Samane S, Yadollah ZP, Marzieh H, Karimollah HT, Reza ZM, Afsaneh A, Als H. Cue-based feeding and short-term health outcomes of premature infants in newborn intensive care units: a non-randomized trial. BMC Pediatr. 2022 Jan 6;22(1):23. doi: 10.1186/s12887-021-03077-1. PMID 34991513
- [Background] Pineda R, Harris R, Foci F, Roussin J, Wallendorf M. Neonatal Eating Outcome Assessment: tool development and inter-rater reliability. Acta Paediatr. 2018 Mar;107(3):414-424. doi: 10.1111/apa.14128. Epub 2017 Dec 8. PMID 29059481
- [Background] Thoyre SM, Shaker CS, Pridham KF. The early feeding skills assessment for preterm infants. Neonatal Netw. 2005 May-Jun;24(3):7-16. doi: 10.1891/0730-0832.24.3.7. PMID 15960007
- [Background] Lubbe W. Clinicians guide for cue-based transition to oral feeding in preterm infants: An easy-to-use clinical guide. J Eval Clin Pract. 2018 Feb;24(1):80-88. doi: 10.1111/jep.12721. Epub 2017 Mar 2. PMID 28251754
- [Background] Crapnell TL, Rogers CE, Neil JJ, Inder TE, Woodward LJ, Pineda RG. Factors associated with feeding difficulties in the very preterm infant. Acta Paediatr. 2013 Dec;102(12):e539-45. doi: 10.1111/apa.12393. Epub 2013 Sep 30. PMID 23952198
- [Background] Adams-Chapman I, Bann CM, Vaucher YE, Stoll BJ; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Association between feeding difficulties and language delay in preterm infants using Bayley Scales of Infant Development-Third Edition. J Pediatr. 2013 Sep;163(3):680-5.e1-3. doi: 10.1016/j.jpeds.2013.03.006. Epub 2013 Apr 10. PMID 23582139
- [Background] Goday PS, Huh SY, Silverman A, Lukens CT, Dodrill P, Cohen SS, Delaney AL, Feuling MB, Noel RJ, Gisel E, Kenzer A, Kessler DB, Kraus de Camargo O, Browne J, Phalen JA. Pediatric Feeding Disorder: Consensus Definition and Conceptual Framework. J Pediatr Gastroenterol Nutr. 2019 Jan;68(1):124-129. doi: 10.1097/MPG.0000000000002188. PMID 30358739
- [Background] Alshaikh B, Yusuf K, Dressler-Mund D, Mehrem AA, Augustine S, Bodani J, Yoon E, Shah P; Canadian Neonatal Network (CNN) and Canadian Preterm Birth Network (CPTBN) Investigators. Rates and Determinants of Home Nasogastric Tube Feeding in Infants Born Very Preterm. J Pediatr. 2022 Jul;246:26-33.e2. doi: 10.1016/j.jpeds.2022.03.012. Epub 2022 Mar 14. PMID 35301017
- [Background] Macias R, Peterson D, Korkis L, Edson R, Gall R. Prevalence and Impact of Feeding-Related Events on Hospital Stay in Preterm and Term Newborns. Adv Neonatal Care. 2023 Dec 1;23(6):541-546. doi: 10.1097/ANC.0000000000001115. Epub 2023 Oct 19. PMID 37862366
- [Background] Hannan KE, Hwang SS, Bourque SL. Readmissions among NICU graduates: Who, when and why? Semin Perinatol. 2020 Jun;44(4):151245. doi: 10.1016/j.semperi.2020.151245. Epub 2020 Mar 13. PMID 32253024
- [Background] Edwards L, Cotten CM, Smith PB, Goldberg R, Saha S, Das A, Laptook AR, Stoll BJ, Bell EF, Carlo WA, D'Angio CT, DeMauro SB, Sanchez PJ, Shankaran S, Van Meurs KP, Vohr BR, Walsh MC, Malcolm WF; Eunice Kennedy Shriver National Institute of Child Health and Human Development. Inadequate oral feeding as a barrier to discharge in moderately preterm infants. J Perinatol. 2019 Sep;39(9):1219-1228. doi: 10.1038/s41372-019-0422-x. Epub 2019 Jul 11. PMID 31296918
- See also: Psychometric Properties of the SMART Feeding Tool — https://clinicaltrials.gov/study/NCT05729828
- See also: Psychometric Properties of SMART Feeding Tool - AHMW SHARE — https://institutionalrepository.aah.org/sciday/2024/oral3/3/